CLINICAL TRIAL: NCT05490095
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetic and Safety After Oral Administration of SVG101(Dispersible Tablet of Everolimus) 5mg and Afinitor 5mg in Healthy Adults
Brief Title: Randomized Crossover of SVG101(Dispersible Tab. of Everolimus) and Afinitor 5mg in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sovargen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SVG101-P1-01
Record Dates: First submitted 2022-08-02; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Pharmacokinetics
Keywords: Everolimus; Healthy adults; Disperse formulation
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): 13 subjects will receive
  1. First Dose: Afinitor 5mg, single dose
  2. Wash out period : more than 10 days
  3. Second Dose: SVG101 5mg, single dose
  Interventions: Drug: SVG101 (T); Drug: Afinitor (R)
- Group II (Experimental): 13 subjects will receive
  1. First Dose: SVG101 5mg, single dose
  2. Wash out period : more than 10 days
  3. Second Dose: Afinitor 5mg, single dose
  Interventions: Drug: SVG101 (T); Drug: Afinitor (R)

INTERVENTIONS:
Drug: SVG101 (T) — 5mg of SVG101
Drug: Afinitor (R) — 5mg of Afinitor

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and safety of SVG101 (dispersible tab. of everolimus) in healthy volunteers compared to Afinitor tab. after oral administration.

DETAILED DESCRIPTION:
This is a randomized, open-label, single-dose, two-way cross-over study to investigate the Pharmacokinetic characteristics and safety after oral administration of SVG101 (dispersible tablet of everolimus) 5mg and Afinitor 5mg in 26 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults: 19y - 55y (Male or Female)
2. Male: more than 55kg, Female: more than 50kg body weight
3. Body mass index: more than 18.5kg/m^2 and less than 27.0kg/m^2
4. Menopause or surgical infertility female

Exclusion Criteria:

1. Participants have or had a history of the clinically relevant disease or abnormalities in the hepatobiliary system, kidney, nervous system, immune system, respiratory system, urinary system, digestive system, endocrine system, blood/tumor, cardiovascular system, and mental illness.
2. Participants with galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
3. Any history of gastrointestinal disease or surgery
4. Participants have hypersensitive to the everolimus or other rapamycin derivatives or other components of the investigational product.
5. Taking any drugs that induce or inhibit metabolizing enzymes such as barbiturate drugs within 30 days prior to first administration
6. Receiving any investigational therapy of others within 180 days prior to first administration. In case of biological products, the restricted period can be extended depend on the half-life receipt product
7. Pregnant or breastfeeding women

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
AUCinf of everolimus | up to 144 hours
Cmax of Everolimus | up to 144 hours
Cmin,ss,pred of Everolimus | up to 144 hours
AUClast of Everolimus | up to 144 hours
Tmax of Everolimus | up to 144 hours
t1/2 of Everolimus | up to 144 hours
Vd/F of Everolimus | up to 144 hours
Clearance of Everolimus | up to 144 hours

SECONDARY OUTCOMES:
Adverse Events (AEs) | up to approximately 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Maeng, Study Director — Sovargen
Locations (1):
- Yonsei University Healthcare System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim JS, Kim WI, Kang HC, Kim SH, Park AH, Park EK, Cho YW, Kim S, Kim HM, Kim JA, Kim J, Rhee H, Kang SG, Kim HD, Kim D, Kim DS, Lee JH. Brain somatic mutations in MTOR cause focal cortical dysplasia type II leading to intractable epilepsy. Nat Med. 2015 Apr;21(4):395-400. doi: 10.1038/nm.3824. Epub 2015 Mar 23. PMID 25799227
- See also: Everolimus_Clinical Pharmacology Review — https://www.accessdata.fda.gov/drugsatfda_docs/nda/2012/203985Orig1s000ClinPharmR.pdf